CLINICAL TRIAL: NCT01991002
Title: Prospective Interventional Study of the Impact of 3-step Diet With Complimentary Exercise Program
Brief Title: 14/21 Diet-walking in the Park
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Principal Investigator, Prof. Sh.Shemer, chairman of the board, Assuta Hospital Systems
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: diet003
Record Dates: First submitted 2013-10-21; First posted 2013-11-25 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Overweight: 25 <BMI <30
Keywords: 14/21 diet; BMI; biochemical blood markers; quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14/21 diet (Other): Diet program is divided into 3 periods: 1. Low carb diet for 14 days; 2. Low carb and regular diet in alternating days for 21 days; 3. Individual carbohydrate-rich diet for 21 days.
  The diet consists of a free choice of food ingredients from a detailed list of foods in each category (proteins, carbohydrates, vegetables, fat etc.). The participants are free to choose the types of food as long as they are within the specified allowance (quantity) for each food group.
  Interventions: Behavioral: 14/21 diet

INTERVENTIONS:
Behavioral: 14/21 diet — Diet program is divided into 3 periods: 1. Low carb diet for 14 days; 2. Low carb and regular diet in alternating days for 21 days; 3. Individual carbohydrate-rich diet for 21 days.
  The diet consists of a free choice of food ingredients from a detailed list of foods in each category (proteins, carbohydrates, vegetables, fat etc.). The participants are free to choose the types of food as long as they are within the specified allowance (quantity) for each food group.

SUMMARY:
The scientific literature shows a quantitative relationship between diet combined with physical activity as a long term weight reduction modality and an important factor in weight maintenance.

Primary assumption - the 14/21 diet will have an impact on BMI values, and their long-term maintenance.

Secondary assumption - the 14/21 diet will have a positive impact on anthropomorphic and biochemical markers, on blood pressure, resting heart rate, RMR, and life quality.

DETAILED DESCRIPTION:
An interventional part for a duration of 56 days and a follow-up period including monitoring of different parameters. Follow up session are set to 3, 6, 12 and 24 months from the end of the interventional period.

Participants will be recruited in several rounds, each including up to 25 participants. Diet program is divided into 3 periods: 1. Low carb diet for 14 days; 2. Low carb and regular diet in alternating days for 21 days; 3. Individual carbohydrate-rich diet for 21 days.

The diet consists of a free choice of food ingredients from a detailed list of foods in each category (proteins, carbohydrates, vegetables, fat etc.). The participants are free to choose the types of food as long as they are within the specified allowance (quantity) for each food group.During the intervention period subjects will meet for walking. In addition, 30 minutes of aerobic exercise will be recommended 3 times/week.

ELIGIBILITY:
Inclusion Criteria:

Hebrew speaking 25<BMI<30 18 years old or older signed an informed consent

Exclusion Criteria:

Subjects who have a physical disability preventing them from exercise, Subjects who are pregnant or lactating, Subjects who are currently involved in another lifestyle intervention program, Subjects who had undergone bariatric surgery in the past, Subjects with: cancer, liver/kidney disease, organ transplantation, alcohol/drug addiction, Subjects that have cognitive deterioration or psychosis, vegetarians who does't eat fish/sea food or vegans

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Weight reduction | 2 years
  BMI will be calculated by the equation weight divided by square height.

SECONDARY OUTCOMES:
Anthropometric measurements | 2 years
  Waist circumference will be measured at the level of the umbilicus. Hip circumference will be measured at the widest portion of the buttocks. Waist/hip ratio will be calculated. "Tanita" will be used for body composition analysis (%fat mass, fat mass,fat free mass and RMR).

OTHER OUTCOMES:
Biochemical markers | 2 years
  To measure glucose, HbA1C (Glycated hemoglobin), blood fat profile, liver enzymes, inflammatory markers.
Blood pressure | 2 years
  Blood pressure will be measured.
Quality of life. | 2 years
  Visual Analog Scale questionnaire and SF-12 questionnaire will be filled out by the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Shemer, Prof., Principal Investigator — Assuta Hospital Systems
Locations (1):
- Assuta medical centers, Tel Aviv, Israel